CLINICAL TRIAL: NCT04130308
Title: Predictive Factors for a Successful Return to Run After Anterior Cruciate Ligament Reconstruction and Underlying Bio-mechanical Factors
Brief Title: Predictive Factors for a Successful Return to Run After ACL-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Ordre Professionnel de la Physiothérapie du Québec (OPPQ) (Unknown)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Associate Professor, Faculty of Medicine, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACLR/Running 2019
Record Dates: First submitted 2019-10-11; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL-R (Experimental)
  Interventions: Other: Retrun to run protocol
- Control (No Intervention)

INTERVENTIONS:
Other: Retrun to run protocol — Progressive return to run protocol for patients after ACL-R
  Arms: ACL-R

SUMMARY:
After anterior cruciate ligament (LCA) rupture, the recommended treatment for athletes is the surgical reconstruction of the ligament (ACL-R), followed by a long rehabilitation period. The results of this treatment are sub-optimal with a low rate of return to pre-injury level of sport, a high risk of reinjury and early knee osteoarthritis. To improve treatment outcomes, researchers and clinicians recommend optimizing rehabilitation protocols. They recommend individualizing rehabilitation progression based on objective criteria. However, current defined criteria relied on experts' opinions and not scientific validation.

Return to run after ACL reconstruction is an important rehabilitation milestone. It often means the beginning of the return to sport continuum. A successful return to run is therefore crucial for both the patient and clinician. In this study, the investigators aim to determine the predictive outcomes for a successful return to run after ACL-R.

ELIGIBILITY:
Experimental group

Inclusion Criteria:

* ACL-R 3 to 4 months ago

Exclusion Criteria:

* already returned to run
* multiple ligament lesions

Control group

Inclusion Criteria:

- healthy person

Exclusion Criteria:

* history of ACL lesion or reconstruction
* history of knee injury
* injured in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Muscular strength assessment | Day 0
  Quadriceps, hamstring and gluteus strength assessment with handheld dynamometer (N)
Modified Y-balance test | Day 0
  Modified Y-balance test (m)
step-down test | Day 0
  endurance test, number of repetition
Self-reported outcomes: ACL-RSI | Day 0
  ACL-RSI: 0-100
Self-reported outcomes: IKDC | Day 0
  IKDC: 0-100

SECONDARY OUTCOMES:
Running kinematic | Day 0 and Day 14
  knee kinematic (degree)
Running kinetic | Day 0 and Day 14
  kinetic (N)
Knee joint contact force | Day 0 and Day 14
  knee joint contact force (N)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, PhD, Principal Investigator — Laval University
Locations (1):
- Center for Interdisciplinary Research in Rehabilitation and Social Integration (CIRRIS), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No